CLINICAL TRIAL: NCT04673552
Title: Open Surgery for Necrotizing Pancreatitis in the Era of Minimally Invasive Approach: 10-year Experience in a High-volume Centre
Brief Title: Open Surgery for Necrotizing Pancreatitis
Status: Completed | Type: Observational
Sponsor: Northern State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: denimsur1974
Record Dates: First submitted 2020-12-12; First posted 2020-12-17 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Pancreatitis,Acute Necrotizing
Keywords: necrotizing pancreatitis; laparotomy; debridement
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing | interventions — Laparotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laparotomy — Any open procedure such as laparotomy or lumbotomy for acute necrotizing pancreatitis will be evaluated, with assessment of results, complications and deaths
  Other Names: lumbotomy; minimally invasive debridement

SUMMARY:
Retrospective analysis of the cases of traditional open surgery for acute necrotizing pancreatitis, with evaluation of indications for surgery, intraoperative findings, mortality rate and risk factors of mortality.

DETAILED DESCRIPTION:
All cases of laparotomy/lumbotomy will be retrospectively analysed, with evaluation of mortality, complications, in-hospital stay, indications for surgery, findings during operation, combination with minimally invasive procedures (radiological drainage, necrosectomy). Assessment of risk factors, like erosive bleeding, intraperitoneal perforation of collection, gut resection, splenectomy, relaparotomy will be done.

ELIGIBILITY:
Inclusion Criteria:

* laparotomy or lumbotomy performed for acute necrotizing pancreatitis from January, 2008 to December, 2017

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-hospital patients of the First Emergency City Hospital named after E. E. Volosevich
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
survival | 01.001.2008 - 31.12.2017
  patient's discharge from the hospital
death | 01.001.2008 - 31.12.2017
  patient's death after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Denis Mizgirev, DoctMedSci, Principal Investigator — Northern State Medical University
Locations (1):
- Northern State Medical University, Arkhangelsk, Arkhangelskaya oblast, Russia

IPD SHARING:
Plan to Share IPD: No